CLINICAL TRIAL: NCT02010463
Title: Neuroimaging Studies of Reward, Impulsivity, and Adherence to an Exercise Program
Brief Title: Neuroimaging Study of Factors Related to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5R01DK085605-04 (NIH); 5R01DK085605 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: reward processing; impulse control; obese; clinically obese
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Intervention (Other): 9-month exercise program involving four exercise education sessions
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
This study aims to support the hypothesis that brain processes underlying reward processing and impulse control contribute to obesity and to adherence in a new exercise regimen.

DETAILED DESCRIPTION:
This is a nonrandomized trial with groups being defined by BMI and adherence status to the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 to < 40±1
* Must live in the Greater Kansas City area for at least 1 year
* Willing to exercise
* Provide written approval from a licensed physician that they are healthy enough to participate in a program of moderate physical activity and maximum O2 testing
* All participants must be sedentary except for casual recreation such as softball, bowling, etc.

Exclusion Criteria:

* Color-blindness
* Left-handedness
* Any diagnosed neurological disorder or conditions that preclude MRI scanning (e.g., metal in body)
* Participation in a research project involving weight loss or physical activity in the previous 6 months
* Subjects who smoke
* Subjects use medications that affect metabolism (i.e. thyroid, beta blockers), use medications that affect appetite (i.e. Meridia) or cannot exercise (i.e. walk)
* Participants will be excluded by study personnel following interview if they exhibit eating disorders, binge eating, depression or drug addiction
* Metabolic disease that would affect energy balance (e.g. diabetes mellitus or hypothyroidism)
* Pregnant during the previous 6 months, are lactating, or plan pregnancy within 12 months
* Individuals who are not weight stable (± 4.5kg) within the previous year.
* Serious medical risks such as type 1-diabetes, cancer, recent cardiac event (i.e. heart attack, angioplasty, etc.)
* High blood pressure
* Current use of smoking/tobacco products or initiation of the use of smoking/tobacco products during the study and alcohol abuse and any history of dependence
* Subject IQ is less that 80
* Reported radiation exposure from CT, PET, fluoroscopic or nuclear medicine studies within the previous year, or other radiation exposure at the discretion of the PI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Body weight and body composition | Change from Baseline to 9 months
  Body weights will be recorded using a digital scale accurate to + 0.1 kg (Befour Inc Model #PS6600, Saukville, WI). Participants will report to the Center between 7 and 10 AM and will be weighed prior to breakfast and after attempting to void. Participants will wear a standard hospital gown at the time of weighing.

SECONDARY OUTCOMES:
Body weight and body composition | Change from Baseline to 4 Months
  Body weights will be recorded using a digital scale accurate to + 0.1 kg (Befour Inc Model #PS6600, Saukville, WI). Participants will report to the Center between 7 and 10 AM and will be weighed prior to breakfast and after attempting to void. Participants will wear a standard hospital gown at the time of weighing.
Treadmill testing for maximum oxygen consumption | Change from Baseline to 4 Months
  Participants will undergo a physician supervised maximal treadmill test to assess changes in maximal oxygen consumption. Furthermore, maximal heart rate obtained from the baseline test will be used to target the appropriate exercise intensity. Participants will walk at 3.4 mph beginning at 0% grade. The grade will be increased 2.5% at 2 minute intervals until exhaustion occurs. Heart rates will be recorded at one minute intervals with a multiple channel electrocardiograph. Expired air will be measured for oxygen and carbon dioxide at 20-second intervals using a ParvoMedics TrueOne 2400 indirect calorimetry system. The system will be and calibrated before each test according to the specifications of the manufacturer (ParvoMedics, Inc Sandy, Utah). Maximal oxygen consumption will be considered as the highest observed value (American College of Sports Medicine 2000).
Treadmill testing for maximum oxygen consumption | Change from Baseline to 9 Months
  Participants will undergo a physician supervised maximal treadmill test to assess changes in maximal oxygen consumption. Furthermore, maximal heart rate obtained from the baseline test will be used to target the appropriate exercise intensity. Participants will walk at 3.4 mph beginning at 0% grade. The grade will be increased 2.5% at 2 minute intervals until exhaustion occurs. Heart rates will be recorded at one minute intervals with a multiple channel electrocardiograph. Expired air will be measured for oxygen and carbon dioxide at 20-second intervals using a ParvoMedics TrueOne 2400 indirect calorimetry system. The system will be and calibrated before each test according to the specifications of the manufacturer (ParvoMedics, Inc Sandy, Utah). Maximal oxygen consumption will be considered as the highest observed value (American College of Sports Medicine 2000).
Measurement of Energy Intake | Change from Baseline to 4 Months
  Participants will be asked not to alter their dietary intake during the intervention. Dietary intake will be documented from 3-day food records (2 weekdays, 1 weekend day). The nutrient content of the record data will be determined using Nutrition Data System for Research (NDS-R, version 2008, University of Minnesota, Minneapolis, MN).
Measurement of Energy Intake | Change from Baseline to 9 Months
  Participants will be asked not to alter their dietary intake during the intervention. Dietary intake will be documented from 3-day food records (2 weekdays, 1 weekend day). The nutrient content of the record data will be determined using Nutrition Data System for Research (NDS-R, version 2008, University of Minnesota, Minneapolis, MN).

CONTACTS AND LOCATIONS:
Overall Officials: Cary Savage, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas, Lawrence, Kansas